CLINICAL TRIAL: NCT03095729
Title: Cognitive Consequences of an Activation of the Cortical Drive to Breath
Brief Title: Cognitive Consequences of an Activation of the Cortical Drive to Breath (VENTIPSY)
Acronym: VENTIPSY
Status: Completed | Type: Observational
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Collaborators: Association Française du Syndrome d'Ondine (Unknown); Fonds de Recherche en Santé Respiratoire (Unknown)
Responsible Party: Sponsor
Other Study IDs: ADOREPS_2017_9
Record Dates: First submitted 2017-03-09; First posted 2017-03-30 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Ondine Syndrome; Healthy; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Sleep Apnea, Central; Amyotrophic Lateral Sclerosis | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy: 40 healthy subjects, during quiet breathing and under an inspiratory load (inspiratory threshold loading)
  Interventions: Other: Neuropsychological tests
- Ondine syndrome: 12 patients presenting with central hypoventilation syndrome or Ondine's curse syndrome, during spontaneous breathing and with Non Invasive Ventilation
  Interventions: Other: Neuropsychological tests
- Amyotrophic Lateral Sclerosis: 30 patients presenting with Amyotrophic Lateral Sclerosis during spontaneous breathing and with Non Invasive Ventilation
  Interventions: Other: Neuropsychological tests

INTERVENTIONS:
Other: Neuropsychological tests — A battery of tests to evaluate the overall cognitive performance of the subjects (memory, executive, attentional or instrumental functions)

SUMMARY:
The purpose of the study is to measure the negative cognitive consequences of the ventilation under pathological or experimental cortical drive to breath.

DETAILED DESCRIPTION:
Cognitive capacities are measured on healthy subject submitted to inspiratory threshold loading, patients treated by chronic mechanical ventilation due to suffering Ondine syndrome or amyotrophic lateral sclerosis. The spontaneous breathing is compared to NIV breathing or inspiratory threshold loading.

ELIGIBILITY:
Inclusion Criteria:

* Adults and non-vulnerable adults
* Fluent in French

Exclusion Criteria:

For patients:

* Total ventilatory dependency
* Coexistence of an other respiratory disease
* Alcohol and /or psychotropic consumption during the last 24 hours
* One or more episodes of acute respiratory failure during the past 6 months
* Serious cognitive deficiency or presence of fronto temporal dementia
* End-stage disease
* No affiliation to social security

For healthy volunteers:

* Existing respiratory disease
* Alcohol and /or psychotropes consumption during the last 24 hours
* Tobacco smoking more than 2 pack-years
* Sleep deprivation
* Serious cognitive deficiency
* No affiliation to social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Score at PASAT (Paced Auditory Serial Addition Test) | 3 hours
  Performances will be assessed by counting the number of good and wrong answers, and comparing it in two conditions : spontaneous breathing (SB) versus inspiratory resistive loading for healthy subjects, and SB versus non invasive ventilation for patients.

SECONDARY OUTCOMES:
Oxygen saturation changes | 3 hours
  Modifications of oxygen saturation measured using a saturometer placed on the subject's finger.

CONTACTS AND LOCATIONS:
Locations (1):
- INSERM-UPC UMR_S 1158, Service de Pneumologie et Réanimation, GH Pitié-Salpêtrière, Paris, France